CLINICAL TRIAL: NCT01841645
Title: Conjugated Linoleic Acid (CLA) Depletion-repletion: Metabolism and Bioactivity in Humans
Brief Title: CLA Metabolism and Effects on Human Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandre Guedes Torres (Other)
Collaborators: Rio de Janeiro State University (Other)
Responsible Party: Sponsor-Investigator, Alexandre Guedes Torres, Professor Alexandre Guedes Torres, Universidade Federal do Rio de Janeiro
Organization: Universidade Federal do Rio de Janeiro (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AGT2013
Record Dates: First submitted 2013-04-17; First posted 2013-04-26 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Dietary Modification; Inflammation; Body Composition, Beneficial
Keywords: CLA-enriched butter; CLA metabolism; inflammation
MeSH Terms: conditions — Inflammation; Glucocorticoid Receptor Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CLA depletion-repletion (Other)
  Interventions: Dietary Supplement: CLA depletion-repletion

INTERVENTIONS:
Dietary Supplement: CLA depletion-repletion

SUMMARY:
The purpose of the study is to investigate the effects of Conjugated Linoleic Acid (CLA) from dairy products on fatty acid metabolism and human health. A CLA depletion-repletion study was carried out with healthy volunteers. CLA depletion was achieved through an eight-week dairy fat restriction, followed by an eight-week repletion period consisting of intake of a butter naturally enriched with CLA. Changes in body composition, fasting glucose and insulin, inflammatory mediators, cell membranes' stability, plasma lipid levels and fatty acid composition of lipid classes are evaluated after depletion and repletion phases.

DETAILED DESCRIPTION:
After collecting baseline blood samples, CLA-depletion phase started with dietary orientation, by a registered dietitian, to the study subjects (n=29) to exclude from their diets any type of dairy fat for the following 8 weeks. Blood samples were taken at the end of CLA-depletion, and CLA-repletion phase was initiated by dietitians' instructions: volunteers returned to their regular diets, and additionally consumed a CLA-enriched butter for another 8-week period. Blood samples were taken at the end of the CLA-repletion phase. The effects of CLA on the following parameters were evaluated: inflammatory mediators; fatty acid composition of erythrocytes, plasma phospholipids and cholesterol esters; body composition; clinical factors associated with the metabolic syndrome and indicators of cell membranes' stability.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers;
* 20 to 40 years;
* BMI between 18.0 and 29.9 kg/m2.

Exclusion Criteria:

* Use of dietary supplements;
* Smoker;
* Alcoholic;
* Under medication;
* History of chronic disease

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2009-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Fatty acid metabolism and inflammatory mediators were accompanied during a CLA depletion-repletion dietary intervention | 16 weeks
  Changes in body composition, fasting glucose and insulin, inflammatory mediators, cell membrane stability, plasma lipid levels and fatty acid composition of lipid classes were evaluated before and after depletion and repletion phases.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre G Torres, DSc, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Federal University of Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil